CLINICAL TRIAL: NCT03320200
Title: A Central Nervous System Focused Treatment Approach for People With Frozen Shoulder: Protocol for a Randomised Clinical Trial
Brief Title: A Central Nervous System Focused Treatment Approach for Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Enrique Lluch Girbés, PhD Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H1507114540624
Record Dates: First submitted 2017-10-12; First posted 2017-10-25 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Adhesive Capsulitis of Shoulder; Frozen Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CNS-focused treatment (Experimental): Group of subjects receiving a 10 week CNS (Central Nervous System) -focused treatment program for frozen shoulder in addition to 5 days per week home treatment program
  Interventions: Other: CNS-focused treatment
- Standard Care Treatment (Experimental): Group of subjects receiving a 10 week standard care treatment program for frozen shoulder in addition to 5 days per week home treatment program based on conventional physiotherapy
  Interventions: Other: Standard Care Treatment

INTERVENTIONS:
Other: CNS-focused treatment — The CNS-focused treatment will last for 10 weeks, conducted in 60-minute sessions on a weekly basis. In addition, participants in this group will complete a home treatment program for 30 minutes, five times a week.
  Other Names: graded motor and sensory imagery traininng
  Arms: CNS-focused treatment
Other: Standard Care Treatment — The standard physiotherapy group will receive a 10-session treatment program that will include one corticosteroid infiltration provided in the early acute stage followed by a multimodal physiotherapy program including analgesic modalities (e.g. TENS, cryotherapy) and exercise and manual therapy techniques addressing the specific mobility deficits of each patient. This program also include a home treatment based on conventional physiotherapy that involves a training load comparable to that in the CNS-focused group.
  Other Names: Conventional physiotherapy treatment
  Arms: Standard Care Treatment

SUMMARY:
The aim of this study is to compare the effectiveness of a CNS-directed treatment program versus a standard medical and physiotherapy care program on outcomes in participants with FS.Participants will be randomized to receive either a 10 weeks CNS-focused treatment program or standard medical and physiotherapy care.To evaluate the results of the interventions, the subjects will be assessed at the beginning, at the end of the treatment program (week 10) and at 3 and 6 months of follow-up.

DETAILED DESCRIPTION:
The aim of this study is to compare the effectiveness of a CNS-directed treatment program versus a standard medical and physiotherapy care program on outcomes in participants with Frozen Shoulder (FS). It will consist of a randomized double-blind clinical trial (both participants and evaluators). The sample will consist of subjects with primary or idiopathic FS.

Once the sample is selected, participants will be randomly assigned to receive either a CNS-centered treatment program or a standard physiotherapy program. The CNS-centered treatment program will last for 10 weeks, conducted in 60-minute sessions on a weekly basis. In addition, participants in this group will complete a home treatment program for 30 minutes, five times a week. On the other hand, subjects assigned to the standard physiotherapy group will receive a 10-session treatment program, such as the CNS-centered treatment group. This standard treatment will include one corticosteroid infiltration provided in the early acute stage followed by a multimodal physiotherapy program including analgesic modalities (e.g. TENS, cryotherapy) and exercise and manual therapy techniques addressing the specific mobility deficits of each patient. Physiotherapists will be instructed not to include interventions that were similar to those used in the group receiving the CNS-focused protocol (e.g. using mirrors or imagined movements) and to include a home program that involves a training load comparable to that in the other group. Adherence to both interventions will be monitored using an individual treatment diary where the time of day and duration of each clinic and home session will be recorded To evaluate the results of the interventions, the subjects will be assessed at the beginning, at the end of the treatment program (week 10) and at 3 and 6 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Primary or idiopathic Frozen Shoulder (FS), defined as FS not associated with a systemic condition or history of injury
* greater than 50% reduction in passive external rotation when compared to the uninvolved shoulder or less than 30° of external rotation
* range of motion loss of greater than 25% in at least two movement planes in comparison to the uninvolved shoulder
* pain and restricted movement present for at least one month reaching a plateau or worsening
* normal shoulder X-rays (with the exception of osteopenia of the humeral head and calcific tendinosis)

Exclusion Criteria:

* Locked dislocations, arthritis, fractures or avascular necrosis on radiographs
* surgery in the upper quadrant region <12 months prior to the study
* skin or medical conditions that prevents from receiving tactile stimuli on the shoulder
* neurological or motor disorders including a diagnosis of dyslexia or difficulty performing a rapid naming task
* visually and mental health conditions that precludes successful participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
shoulder pain-related disability questionnaire (SPADI) | Baseline
  The SPADI is a 13-items shoulder function index assessing pain and disability related to shoulder dysfunction. Each item is scored by a numeric rate scale ranging from 0 (no pain/no difficulty) to 10 (worst pain imaginable/so difficult it required help). The total score ranges from 0 to 100 points where a higher score indicates greater disability.
shoulder pain-related disability questionnaire (SPADI) | Change from baseline SPADI at 10 weeks
  The SPADI is a 13-items shoulder function index assessing pain and disability related to shoulder dysfunction. Each item is scored by a numeric rate scale ranging from 0 (no pain/no difficulty) to 10 (worst pain imaginable/so difficult it required help). The total score ranges from 0 to 100 points where a higher score indicates greater disability.
shoulder pain-related disability questionnaire (SPADI) | Change from baseline SPADI at 3 months
  The SPADI is a 13-items shoulder function index assessing pain and disability related to shoulder dysfunction. Each item is scored by a numeric rate scale ranging from 0 (no pain/no difficulty) to 10 (worst pain imaginable/so difficult it required help). The total score ranges from 0 to 100 points where a higher score indicates greater disability.
shoulder pain-related disability questionnaire (SPADI) | Change from baseline SPADI at 6 months
  The SPADI is a 13-items shoulder function index assessing pain and disability related to shoulder dysfunction. Each item is scored by a numeric rate scale ranging from 0 (no pain/no difficulty) to 10 (worst pain imaginable/so difficult it required help). The total score ranges from 0 to 100 points where a higher score indicates greater disability.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | Baseline
  a valid and reliable measure of shoulder pain. Participants will be presented with numerical rating scales anchored with 0 ("no pain") and 10 ("pain as bad as you can imagine").
Numeric Pain Rating Scale | Change from baseline Numeric Rating Pain Scale at 10 weeks
  a valid and reliable measure of shoulder pain. Participants will be presented with numerical rating scales anchored with 0 ("no pain") and 10 ("pain as bad as you can imagine").
Numeric Pain Rating Scale | Change from baseline Numeric Rating Pain Scale at 3 months
  a valid and reliable measure of shoulder pain. Participants will be presented with numerical rating scales anchored with 0 ("no pain") and 10 ("pain as bad as you can imagine").
Numeric Pain Rating Scale | Change from baseline Numeric Rating Pain Scale at 6 months
  a valid and reliable measure of shoulder pain. Participants will be presented with numerical rating scales anchored with 0 ("no pain") and 10 ("pain as bad as you can imagine").
Goniometric assessment of active shoulder ROM (range of motion) | Baseline
  Degrees of active range of motion
Goniometric assessment of active shoulder ROM (range of motion) | Change from baseline ROM at 10 weeks
  Degrees of active range of motion
Goniometric assessment of active shoulder ROM (range of motion) | Change from baseline ROM at 3 months
  Degrees of active range of motion
Goniometric assessment of active shoulder ROM (range of motion) | Change from baseline ROM at 6 months
  Degrees of active range of motion
Two point discrimination threshold | Baseline
  Two point discrimination threshold measured at one standardize site on the affected shoulder (5cm distal to the lateral border of the acromion) 33, following an established protocol
Two point discrimination threshold | Change from baseline two point discrimination threshold at 10 weeks
  Two point discrimination threshold measured at one standardize site on the affected shoulder (5cm distal to the lateral border of the acromion) 33, following an established protocol
Two point discrimination threshold | Change from baseline two point discrimination threshold at 3 months
  Two point discrimination threshold measured at one standardize site on the affected shoulder (5cm distal to the lateral border of the acromion) 33, following an established protocol
Two point discrimination threshold | Change from baseline two point discrimination threshold at 6 months
  Two point discrimination threshold measured at one standardize site on the affected shoulder (5cm distal to the lateral border of the acromion) 33, following an established protocol
Laterality judgement accuracy | Baseline
  Laterality judgement accuracy using the NOI Recognise online program (www.noigroup.com) and following and established protocol
Laterality judgement accuracy | Change from baseline laterality judgement accuracy at 10 weeks
  Laterality judgement accuracy using the NOI Recognise online program (www.noigroup.com) and following and established protocol
Laterality judgement accuracy | Change from baseline laterality judgement accuracy at 3 months
  Laterality judgement accuracy using the NOI Recognise online program (www.noigroup.com) and following and established protocol
Laterality judgement accuracy | Change from baseline laterality judgement accuracy at 6 months
  Laterality judgement accuracy using the NOI Recognise online program (www.noigroup.com) and following and established protocol
The Spanish version of the Tampa Scale of Kinesophobia (TSK-11) | Baseline
  The TSK-11 is an 11-item questionnaire assessing fear of movement or fear of (re)injury during movement. It is comprised of 11 items each ranged on a 4-point scale with the end points (1) "totally agree" and (4) "totally disagree" (range: 11-44). Higher scores indicate more fear-avoidance behavior.
The Spanish version of the Tampa Scale of Kinesophobia | Change from baseline Tampa Scale of Kinesophobia at 10 weeks
  The TSK-11 is an 11-item questionnaire assessing fear of movement or fear of (re)injury during movement. It is comprised of 11 items each ranged on a 4-point scale with the end points (1) "totally agree" and (4) "totally disagree" (range: 11-44). Higher scores indicate more fear-avoidance behavior.
The Spanish version of the Tampa Scale of Kinesophobia | Change from baseline Tampa Scale of Kinesophobia at 3 months
  The TSK-11 is an 11-item questionnaire assessing fear of movement or fear of (re)injury during movement. It is comprised of 11 items each ranged on a 4-point scale with the end points (1) "totally agree" and (4) "totally disagree" (range: 11-44). Higher scores indicate more fear-avoidance behavior.
The Spanish version of the Tampa Scale of Kinesophobia | Change from baseline Tampa Scale of Kinesophobia at 6 months
  The TSK-11 is an 11-item questionnaire assessing fear of movement or fear of (re)injury during movement. It is comprised of 11 items each ranged on a 4-point scale with the end points (1) "totally agree" and (4) "totally disagree" (range: 11-44). Higher scores indicate more fear-avoidance behavior.
The Patient Specific Functional Scale | Baseline
  A list of activities and movements is shown to the patients and they are asked to identify the activities that he/she experience difficulty with because of his/her complaints in the shoulder. The patient selects the 3 most important activities and rank them by degree of importance from 0 (no difficulty at all) to 10 (impossible). The total score range from 0 to 30. Higher score indicates higher difficulty in performance on daily activities.
The Patient Specific Functional Scale | Change from baseline Patient Specific Functional Scale at 10 weeks
  A list of activities and movements is shown to the patients and they are asked to identify the activities that he/she experience difficulty with because of his/her complaints in the shoulder. The patient selects the 3 most important activities and rank them by degree of importance from 0 (no difficulty at all) to 10 (impossible). The total score range from 0 to 30. Higher score indicates higher difficulty in performance on daily activities.
The Patient Specific Functional Scale | Change from baseline Patient Specific Functional Scale at 3 months
  A list of activities and movements is shown to the patients and they are asked to identify the activities that he/she experience difficulty with because of his/her complaints in the shoulder. The patient selects the 3 most important activities and rank them by degree of importance from 0 (no difficulty at all) to 10 (impossible). The total score range from 0 to 30. Higher score indicates higher difficulty in performance on daily activities.
The Patient Specific Functional Scale | Change from baseline Patient Specific Functional Scale at 6 months
  A list of activities and movements is shown to the patients and they are asked to identify the activities that he/she experience difficulty with because of his/her complaints in the shoulder. The patient selects the 3 most important activities and rank them by degree of importance from 0 (no difficulty at all) to 10 (impossible). The total score range from 0 to 30. Higher score indicates higher difficulty in performance on daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Lluch, PhD, Study Director — Physiotherapy Department University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

REFERENCES:
- [Result] Wand BM, O'Connell NE, Di Pietro F, Bulsara M. Managing chronic nonspecific low back pain with a sensorimotor retraining approach: exploratory multiple-baseline study of 3 participants. Phys Ther. 2011 Apr;91(4):535-46. doi: 10.2522/ptj.20100150. Epub 2011 Feb 24. PMID 21350034
- [Result] Louw A, Puentedura EJ, Reese D, Parker P, Miller T, Mintken PE. Immediate Effects of Mirror Therapy in Patients With Shoulder Pain and Decreased Range of Motion. Arch Phys Med Rehabil. 2017 Oct;98(10):1941-1947. doi: 10.1016/j.apmr.2017.03.031. Epub 2017 May 5. PMID 28483657
- [Result] Moseley GL. Do training diaries affect and reflect adherence to home programs? Arthritis Rheum. 2006 Aug 15;55(4):662-4. doi: 10.1002/art.22086. No abstract available. PMID 16874790
- [Result] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Result] Moseley G, Butler D, Beames T, Giles T. The graded motor imagery handbook. Adelaide: Noigroup Publishing; 2012.
- [Result] Desroches G, Desmeules F, Gagnon DH. Characterization of humeral head displacements during dynamic glenohumeral neuromuscular control exercises using quantitative ultrasound imaging: A feasibility study. Musculoskelet Sci Pract. 2017 Jun;29:150-154. doi: 10.1016/j.msksp.2016.12.004. Epub 2016 Dec 11. PMID 28715302
- [Result] Mottram SL, Woledge RC, Morrissey D. Motion analysis study of a scapular orientation exercise and subjects' ability to learn the exercise. Man Ther. 2009 Feb;14(1):13-8. doi: 10.1016/j.math.2007.07.008. Epub 2007 Oct 1. PMID 17910930
- [Derived] Mena-Del Horno S, Balasch-Bernat M, Duenas L, Reis F, Louw A, Lluch E. Laterality judgement and tactile acuity in patients with frozen shoulder: A cross-sectional study. Musculoskelet Sci Pract. 2020 Jun;47:102136. doi: 10.1016/j.msksp.2020.102136. Epub 2020 Feb 24. PMID 32148332
- [Derived] Lluch-Girbes E, Duenas L, Mena-Del Horno S, Luque-Suarez A, Navarro-Ledesma S, Louw A. A central nervous system-focused treatment approach for people with frozen shoulder: protocol for a randomized clinical trial. Trials. 2019 Aug 13;20(1):498. doi: 10.1186/s13063-019-3585-z. PMID 31409380